CLINICAL TRIAL: NCT02809664
Title: Feasibility and Safety of Ultrasound Guided Installation Central Subclavian Catheter Through Supraclavicular Way
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6287
Record Dates: First submitted 2016-01-04; First posted 2016-06-22 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Heart Diseases; Diseases, Metabolic
MeSH Terms: conditions — Heart Diseases; Metabolic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Our goal is to demonstrate the feasibility of laying uncomplicated ultrasound-guided central subclavian catheter by supraclavicular route in the newborn.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized in the neonatal intensive care or neonatal intensive care at the University Hospital of Hautepierre
* All infants less than 44 weeks corrected age who require a surgical approach
* In the first line if neonate over 34 weeks corrected age requiring dual carriageway catheter
* After Failure or inability laying KTEC for children between 30 and 34 weeks of age corrected and heavy over 1000

Exclusion Criteria:

* Nouveau-né de poids < 1000g
* Nouveau-né de moins de 30 semaines d'âge corrigé
* Choix d'une autre voie d'abord plus judicieux (KTVO, KTC broviac)
* Sortie avant retrait du KTC

Ages: 43 Weeks to 44 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients hospitalized in the neonatal intensive care or neonatal intensive care.
  The 3 types of taken most often encountered load are:
  1. support for prematurity at birth or poor adaptation at birth requiring intensive care or ventilatory support.
  2. management of congenital heart diseases including ducto-dependent, awaiting surgery.
  3. care for severe medical condition exposing one or more organ failure, between 0 and 28 days of life (severe infections, metabolic diseases, severe dehydration ...)
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2015-10-14 (Actual); Primary Completion 2017-10-14 (Estimated); Study Completion 2017-11-14 (Estimated)

PRIMARY OUTCOMES:
success rate without complications laying catheter ultrasound guided subclavian by supraclavicular route in newborn | 1h after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Kuhn, MD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- Service de réanimation néonatale - HOPITAL DE HAUTEPIERRE, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No